CLINICAL TRIAL: NCT01862718
Title: Fusion Guided Thermal Ablation Combined With External Beam Radiation for Hepatic Neoplasms
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow/Insufficient accrual
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130079; 13-CC-0079
Record Dates: First submitted 2013-05-23; First posted 2013-05-24 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Liver Neoplasms; Hepatic Cancer; Liver Cancer
Keywords: Fusion; Tracking; Ablation; Hepatic Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Ablation plus radiation
  Interventions: Procedure: Thermal Ablation; Procedure: Standard External Beam Radiation Therapy

INTERVENTIONS:
Procedure: Thermal Ablation — On Thursday in the first week, subject will receive the radiofrequency ablation.
Procedure: Standard External Beam Radiation Therapy — During those 2 weeks, subject will receive radiation on Monday, Wednesday and Friday.

SUMMARY:
Background:

Pilot study to assess feasibility for combining treatment modalities that should be synergistic (radiation and thermal ablation).

Thermal ablation with Radiofrequency Ablation (RFA) and microwave ablation (MWA) are standard treatments for focal neoplasms in the liver.

High volume or scattered locations of tumor burden results in inability to successfully use this technology for a large proportion of patients with hepatic neoplasms.

Methods to enhance treatment volumes could be advantageous in potentially increasing the indications for thermal ablation or the number of patients benefitting from local ablation.

Primary objective:

To determine the safety of combining 2 standard therapies (thermal ablation and external beam radiation therapy) for liver neoplasms up to 10 cm diameter.

Eligibility:

Patients greater than 18 years of age with pathologically proven unresectable primary or metastatic hepatic neoplasms

Patients whose extent of hepatic metastases represents approximately less than 60% of total liver volume AND whose extrahepatic metastatic disease is determined to be minimal

ECOG performance status of less than or equal to 2 and a life expectancy of more than 3 months

Patients with a history of chemotherapy, radiation therapy, or biological therapy for at least 4 weeks prior to starting study treatments, and 4 weeks after treatments Patients must not have an acute, critical illness

If clinical or imaging evidence for cirrhosis present, then Bilirubin must be less than 3 mg/dl and Child-Pugh Classification A, (Class B & C are excluded)

Design:

Patients will undergo external beam radiation as well as thermal ablation according to standard operating procedures of the NCI and NIH CC.

Patients will be monitored using the standard imaging studies when clinically warranted.

Patients may be treated with a second (or more) thermal ablation procedure ALONE if it is deemed beneficial for the patient by the investigator.

The sample size will be 10 evaluable patients

DETAILED DESCRIPTION:
Background:

Pilot study to assess feasibility for combining treatment modalities that should be synergistic (radiation and thermal ablation).

Thermal ablation with Radiofrequency Ablation (RFA) and microwave ablation (MWA) are standard treatments for focal neoplasms in the liver.

High volume or scattered locations of tumor burden results in inability to successfully use this technology for a large proportion of patients with hepatic neoplasms.

Methods to enhance treatment volumes could be advantageous in potentially increasing the indications for thermal ablation or the number of patients benefitting from local ablation.

Primary objective:

To determine the safety of combining 2 standard therapies (thermal ablation and external beam radiation therapy) for liver neoplasms up to 10 cm diameter.

Eligibility:

Patients greater than 18 years of age with pathologically proven unresectable primary or metastatic hepatic neoplasms

Patients whose extent of hepatic neoplasms represents approximately less than 60% of total liver volume AND whose extrahepatic metastatic disease is determined to be minimal

ECOG performance status of less than or equal to 2 and a life expectancy of more than 3 months

Patients with a history of chemotherapy, radiation therapy to liver, or biological therapy must have had last dose/ treatment for at least 14 days prior to starting study treatments.

Patients must not have an acute, critical illness

Design:

Patients will undergo external beam radiation as well as thermal ablation according to standard operating procedures of the NCI and NIH CC.

Patients will be monitored using the standard imaging studies when clinically warranted.

Patients may be treated with a second (or more) thermal ablation procedure ALONE if it is deemed beneficial for the patient by the investigator.

The sample size will be 10 evaluable patients

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with hepatic-dominant neoplasms where the life limiting component of the disease is hepatic neoplasms

Patients hepatic lesions must be considered technically unresectable or that their overall health makes surgery inadvisable

Have 5 or fewer lesions and with no single lesion greater than 10 cm in maximum diameter

Patients with extrahepatic neoplasms or an unresected primary lesion will be considered eligible if the extrahepatic disease is minimal and stable

Serum Creatinine less than or equal to 2.0 mg/dl unless the measured creatinine clearance is greater than 60 ml/min.

Absolute neutrophil count (ANC) greater than or equal to1500/m3 without help of Filgastim, hemoglobin greater than 8 g/dL, and platelet count greater than or equal to 75,000 m3

Bilirubin less than 3 mg/dl, and AST and ALT less than 5 X upper limit of normal except in the presence of obstructive liver neoplasms where ALT/AST may be up to 10 X the upper limit of normal.

Prothrombin Time (PT) within 2 seconds of the upper limit normal (INR less than or equal to 1.5)

Patient on oral, SQ or IV anticoagulants will be expected to have an abnormal PT and will be considered eligible if they can safely dicontinue the anticoagulant before ablation. A repeat PT will be obtained at least 24 hours prior to the radiofrequency ablation (only) and should be within practice safety guidelines of an INR less than 1.5 or if greater than 1.5 have clinical reversal agent as appropriate to the anticoagulant administered.

Extent of hepatic neoplasms is approximately less than 60% of total hepatic volume

Patients must have pathology proof of neoplasm. If proof of pathology is unavailable, histopathological confirmation of liver neoplasm may not be requisite in the setting of clinical or radiological characteristics that are highly suggestive of a neoplastic diagnosis, with such designation determined by PI and a medical or surgical oncologist, with the NCI multidisciplinary gastrointestinal tumor board review, in the event of absence of such consensus.

Patients referred for ablation or radiation of liver neoplasm

ECOG performance status less than or equal to 2

Life expectancy greater than 3 months

At least 18 years of age

Age less than 85 years

Patients must have had no chemotherapy, radiotherapy, or biologic therapy for their malignancy for at least 28 days prior to treatment and must have recovered from all clinically significant side effects of therapeutic and diagnostic interventions.

EXCLUSION CRITERIA:

Portal Vein Occlusion or other contraindications to thermal ablation or radiation Prior selective internal radiation therapy (SIRT) with Yttrium-90 or prior radiation to the liver

Prior biliary diversion surgery

Patients with active bacterial infections with systemic manifestations (malaise, fever, leukocytosis) are not eligible until completion of appropriate therapy.

Any exclusion criteria for radiation or for ablation, such as ataxia telangiectasia, active connective tissue disease, or inflammatory bowel disease, or other known conditions which predispose to radiation toxicities

Patients with an acute, critical illness

Pregnant women are excluded from the study. Patients are excluded from pregnancy testing if they are above the childbearing age of 55 years old, or if they have documented history of infertility or acquired or congenital disorders incompatible with pregnancy or if the patient has had a hysterectomy or bilateral oophorectomy. Patients are also excluded from pregnancy testing if they are at least 50 years of age AND have not menstruated for at least 12 months OR have a documented Follicle Stimulating Hormone (FSH) level of greater than 40 mIU/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Safety of Ablation plus radiation | 3 years
  Descriptive statistics will be provided in summary tables. When relevant, the 95% confidence intervals (CI) will also be displayed.

CONTACTS AND LOCATIONS:
Overall Officials: Bradford J Wood, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Background] Komorizono Y, Oketani M, Sako K, Yamasaki N, Shibatou T, Maeda M, Kohara K, Shigenobu S, Ishibashi K, Arima T. Risk factors for local recurrence of small hepatocellular carcinoma tumors after a single session, single application of percutaneous radiofrequency ablation. Cancer. 2003 Mar 1;97(5):1253-62. doi: 10.1002/cncr.11168. PMID 12599233
- [Background] Siperstein AE, Rogers SJ, Hansen PD, Gitomirsky A. Laparoscopic thermal ablation of hepatic neuroendocrine tumor metastases. Surgery. 1997 Dec;122(6):1147-54; discussion 1154-5. doi: 10.1016/s0039-6060(97)90221-x. PMID 9426432
- [Background] Buscarini L, Rossi S, Fornari F, Di Stasi M, Buscarini E. Laparoscopic ablation of liver adenoma by radiofrequency electrocauthery. Gastrointest Endosc. 1995 Jan;41(1):68-70. doi: 10.1016/s0016-5107(95)70279-2. No abstract available. PMID 7698628
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-CC-0079.html